CLINICAL TRIAL: NCT04777058
Title: Pharmacokinetics of Isavuconazole (Cresemba®) Given as Treatment of Invasive Fungal Infections in Patients in the Intensive Care Unit
Brief Title: Pharmacokinetics of Isavuconazole in Patients in the Intensive Care Unit
Acronym: ICONIC
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN-AKF-21.02
Record Dates: First submitted 2021-02-11; First posted 2021-03-02 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Invasive Fungal Infections; Pharmacokinetics; Intensive Care Unit
Keywords: isavuconazole; population pharmacokinetics; protein binding
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood will be obtained and processed to obtain plasma. Plasma levels of total and unbound isavuconazole will be determined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients admitted to the intensive care unit, treated with isavuconazole intravenously for treatment of invasive fungal infections

SUMMARY:
20 patients admitted to the ICU department and receiving isavuconazole as part of standard care for the treatment of fungal infections will be included in the study. Between day 3 and 7, 8 samples will be collected at t = 0 (pre-dose), and t = 0.5, 1, 2, 4, 6, 8 and 12 hours after end of infusion to obtain a PK curve. An optional, additional sample can be collected after discontinuation of isavuconazole therapy if possible. Total and free isavuconazole concentrations will be determined. A pharmacokinetic model will be fitted to the data from all individuals simultaneously. Data will be analysed using non-linear mixed effects modelling (NONMEM).

DETAILED DESCRIPTION:
Fungal infections are a serious threat to immunocompromised patients and represent a major burden in the critical care setting. The azole antifungal drugs are the most important drugs for managing infections caused by Aspergillus moulds and the prevention of invasive fungal infections in general. Azoles are currently used as first line prophylaxis and treatment of invasive aspergillosis and their use has substantially improved the survival of the overall population. Recently, there has been increased awareness for invasive aspergillosis cases in critically ill patients, including patients with severe influenza (influenza associated pulmonary aspergillosis, IAPA), and recently COVID-19 associated pulmonary aspergillosis (CAPA). These patients require azole-based therapy, for which voriconazole and isavuconazole are recommended first choice drugs.

Isavuconazole is a relatively novel azole drug with promising efficacy, a broad antifungal spectrum, favourable side effect profile and limited drug-drug interactions compared to other azole agents. Isavuconazole is registered for the primary treatment of adults with invasive aspergillosis, and patients with mucormycosis where amphotericin B is not suitable. Efficacy and safety information in the isavuconazole label is mostly derived from clinical studies in healthy volunteers. However, the pharmacokinetics in some specific patient populations may differ greatly from those in the healthy population. Changes in pharmacokinetics of isavuconazole in ICU patients are to be expected due to a wide variety of factors, e.g. changes in protein binding and changes in fluid distribution. Therefore, it is likely that the present standard dosing regimens of isavuconazole lead to suboptimal outcomes for ICU patients, similar to observations made for fluconazole and echinocandins. Optimizing dosing regimens in ICU patients for existing antifungal agents such as isavuconazole is important to improve clinical outcome rates. To date, limited information on the pharmacokinetics of isavuconazole in critically ill patients is available and optimal dosing regimens remain uncertain. With this study we aim to describe isavuconazole pharmacokinetics in ICU admitted patients.

20 patients admitted to the ICU department and receiving isavuconazole as part of standard care for the treatment of fungal infections will be included in the study. Between day 3 and 7, 8 samples will be collected at t = 0 (pre-dose), and t = 0.5, 1, 2, 4, 6, 8 and 12 hours after end of infusion to obtain a PK curve. An optional, additional sample can be collected after discontinuation of isavuconazole therapy if possible. Total and free isavuconazole concentrations will be determined. A pharmacokinetic model will be fitted to the data from all individuals simultaneously. Data will be analysed using non-linear mixed effects modelling (NONMEM). NONMEM is a one-stage analysis that simultaneously estimates mean parameters, fixed effect parameters, interindividual variability, and residual random effects. Since allowance can be made for individual differences, this method can be used with both intensive sampling and sparse data (and in the occasion of missing values: an unbalanced number of data points per patients).

Primary objective:

• To determine the pharmacokinetics of isavuconazole given as treatment of invasive fungal infections in ICU patients as part of standard care.

Secondary objectives:

* To investigate the protein binding of isavuconazole in ICU patients and the variability in protein binding between patients in the ICU population.
* To explore if unbound isavuconazole concentrations can be predicted from total isavuconazole concentrations.
* To assess pharmacokinetic/pharmacodynamic target attainment in the ICU patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patient is admitted to an ICU
* Is treated with isavuconazole intravenously (iv)
* Subject is at least 18 years on the day of the first dosing
* Is managed with a central venous catheter or arterial line

Exclusion Criteria:

* Patient has previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty ICU patients treated with isavuconazole for a fungal infection are eligible for inclusion. These patients are admitted to the ICU of Radboudumc and UZ Leuven. Since the objective is to evaluate the pharmacokinetics of isavuconazole in a real-life cohort of patients admitted to the ICU, exclusion criteria are minimal on purpose, to give a good reflection of this heterogenic cohort. The possible inclusion of patients with for example hepatic insufficiencies, continuous renal replacement therapy (CRRT), extracorporeal membrane oxygenation (ECMO) et cetera, is considered. High variability between subjects in this highly heterogenetic patient population is expected and will be considered in the analyses.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Isavuconazole clearance in ICU patients. | Day 3-7 after start of treatment and optional: 96-300 hours after discontinuation of treatment
  Isavuconazole clearance in ICU patients in liters/hour. Full pharmacokinetic curves will be taken and an optional sample during the elimination phase of isavuconazole.
Isavuconazole volume of distribution in ICU patients | Day 3-7 after start of treatment and optional: 96-300 hours after discontinuation of treatment
  Isavuconazole volume of distribution in ICU patients in liters. Full pharmacokinetic curves will be taken and an optional sample during the elimination phase of isavuconazole.

SECONDARY OUTCOMES:
Isavuconazole proteinbinding in ICU patients. | Day 3-7 after start of treatment and optional: 96-300 hours after discontinuation of treatment
  Isavuconazole proteinbinding in ICU patients described by unbound isavuconazole fraction (fu).
Predictability of unbound isavuconazole concentrations | Day 3-7 after start of treatment and optional: 96-300 hours after discontinuation of treatment
  To compare the predicted and observed unbound isavuconazole concentrations in ICU patients: percentage of deviation from predicted.
Target attainment of isavuconazole in ICU patients | At steady state (day 3-7 after start of treatment)
  Percentage of patients reaching the predetermined adequate PK/PD target (isavuconazole trough concentration in mg/l)

CONTACTS AND LOCATIONS:
Locations (4):
- University Hospitals Leuven, Leuven, Belgium
- Netherlands (3):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Radboud University Medical Centre, Nijmegen
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jansen AME, Mertens B, Spriet I, Verweij PE, Schouten J, Wauters J, Debaveye Y, Ter Heine R, Bruggemann RJM. Population Pharmacokinetics of Total and Unbound Isavuconazole in Critically Ill Patients: Implications for Adaptive Dosing Strategies. Clin Pharmacokinet. 2023 Dec;62(12):1701-1711. doi: 10.1007/s40262-023-01305-8. Epub 2023 Oct 11. PMID 37819503